CLINICAL TRIAL: NCT02165683
Title: Investigation of Propranolol Premedication to Reduce FDG Uptake in Brown Adipose Tissue on PET Scans of Pediatric Cancer Patients
Brief Title: Use of Propranolol to Reduce FDG Uptake in Brown Adipose Tissue in Pediatric Cancer Patients PET Scans
Status: Completed | Type: Observational
Sponsor: Lars Wagner (Other)
Responsible Party: Sponsor-Investigator, Lars Wagner, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 14-0468-F3r
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Pediatric Cancer
Keywords: Cancer; Pediatric; PET Scan
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a single-arm, open-label study to assess the safety and effectiveness of a single dose of oral propranolol in reducing18F-fluorodeoxyglucose (FDG) uptake in brown adipose tissue (BAT) in pediatric oncology patients. This study is designed to better understand if taking a single dose of an oral medication called propranolol can reduce the chance of brown fat showing up on a PET scan, and therefore make the scan more accurate and easy to interpret. All humans have some degree of normal brown fat (called brown adipose tissue), and this normal tissue can sometimes light up on a PET scan. That creates problems because it may be wrongly interpreted by the radiologist as tumor, or it may hide true areas of tumor underneath it. Participants will not be randomized and will receive a single dose of oral propranolol approximately 60 minutes prior to the injection of the FDG tracer. The dose of propranolol will be 20 mg for all participants.

DETAILED DESCRIPTION:
In this study, participants will be assessed in the University of Kentucky DanceBlue Pediatric Hematology/Oncology clinic to confirm they are eligible for the study. This will be done at the time intravenous (iv) access is started, either through an iv placed in the arm or through a port/central line.

All females who are capable of becoming pregnant will then undergo urine pregnancy testing. If it is found that they are pregnant they will not be allowed to be in the study. Participant blood sugar will be checked. When possible, the research blood sample will be collected at a time when routine non-research labs will be collected.

Study eligible participants will then be given a single 20 mg tablet of propranolol to take by mouth and will be escorted by a member of the medical team to the PET scan trailer, where they will be checked in and assessed. Blood sugar level will again be checked by finger stick according to the standard procedure for PET scans.

Vital signs will be assessed by a clinical research nurse at least three times while the participants are at the PET scan trailer, including twice before the scan and once immediately after the scan. The nurse will also assess for any symptoms related to the propranolol. If no problems are noted, participants will be discharged from the PET scan trailer and their tudy participation will end. If any side effects arise from the medication, the pediatric oncologist will be called immediately and appropriate treatment started. The PET scan will be assessed by the radiologist to see whether there is uptake in brown fat, as well as to see if any areas of tumor are seen.

ELIGIBILITY:
Inclusion Criteria:

* Individual is between 12 years and 29 years of age
* Individual weighs over 66 pounds
* Individual will be undergoing a FDG-PET scan as part of staging or response assessment for malignancy. Note: the patient may be newly-diagnosed, currently receiving therapy, or have already completed therapy. The presence of identifiable tumor on the PET scan is not required.
* Individual is able to swallow a tablet

Exclusion Criteria:

* Prior diagnosis of asthma, OR use of an inhaler in past three years to treat or prevent bronchospasm.
* History of cardiac arrhythmia requiring treatment
* History of congestive heart failure
* Current use of medications to control blood pressure or improve cardiac output
* Diabetes Type I or II, or currently on medications to reduce blood sugar
* Pregnant

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 11 Male and female participants from all races and ethnic backgrouns who are receiving treatment by the University of Kentucky Medical Center, Pediatric Oncology divsion.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events following Propranolol dosing | 1 day
  The primary objective of our study will be to document the safety of using a single dose of propranolol.

SECONDARY OUTCOMES:
Number of Reductions in FDG Uptake in BATWhen Compared to Historic Controls | 2 years
  We will test the hypothesis that the use of propranolol given prior to the PET scan results in a statistically significant reduction in FDG uptake in BAT compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wagner, MD, Principal Investigator — University of Kentucky, Dept of Pediatric Hematology/Oncology
Locations (1):
- University of Kentucky DanceBlue Pediatric Hematology/Oncology Clinic, Lexington, Kentucky, United States